CLINICAL TRIAL: NCT04241367
Title: Verification of Predictive Biomarkers for Pancreatic Cancer Treatment Using Multicenter Liquid Biopsy
Status: Active, not recruiting | Type: Observational
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Sang Myung Woo, Chief, Senior Scientist, National Cancer Center, Korea
Other Study IDs: NCC2019-0027
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Pancreas Adenocarcinoma
Keywords: Pancreas Adenocarcinoma; Circulating-tumor DNA; KRAS mutations; Cancer Panel; Prognostic markers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study is for verification of predictive biomarkers for pancreatic cancer treatment using multi-center liquid biopsy.

DETAILED DESCRIPTION:
Clinical applicability of KRAS mutations using circulating-tumor DNA in pancreatic cancer patients.

* Quantification and monitoring of KRAS mutations Using droplet digital PCR in ctDNA extracted from collected patient samples.
* Correlation analysis of KRAS mutation results with clinical data.

Discovery of biomarkers for predicting pancreatic cancer prognosis through ctDNA panel.

* Gene panel composition for pancreatic cancer therapeutic target determination and monitoring.
* A panel was performed using gDNA and ctDNA of tumor tissue collected from pancreatic cancer patients.
* Comparative analysis of panel results and quantitative KRAS mutations and evaluation of clinical applicability.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed pancreatic adenocarcinoma.

Exclusion Criteria:

* Patients disagree with the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inpatient or outpatient
Sampling Method: Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical applicability of KRAS mutations | Locally advanced and Resectable patients: Pre Treatment, 1,2,3,6,9,12,15,18,21,24months/ Metastatic patients: Pre Treatment, 1,2,4,6,8,10,12,14,16,18,20,22,24 months
  Clinical applicability of KRAS mutations using circulating-tumor DNA in pancreatic cancer patients.
Discovery of biomarkers through ctDNA panel | Locally advanced and Resectable patients: Pre Treatment, 1,2,3,6,9,12,15,18,21,24months/ Metastatic patients: Pre Treatment, 1,2,4,6,8,10,12,14,16,18,20,22,24 months
  Discovery of biomarkers for predicting pancreatic cancer prognosis through ctDNA panel.

CONTACTS AND LOCATIONS:
Overall Officials: Sangmyung Woo, MD, Principal Investigator — National Cancer Center
Locations (1):
- NATIONAL CANCER CENTER 323, Ilsan-ro, Ilsandong-gu,, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Chun JW, Lee DE, Kim MK, Hwang JH, Lee SH, Jung MK, Kim EJ, Ahn DW, Kim YH, Han SS, Park SJ, Lee WJ, Woo SM, Kong SY. Optimal Value of Mutant KRAS Circulating Tumor DNA for Predicting Prognosis and Monitoring in Patients with Pancreatic Adenocarcinoma: A Prospective Multicenter Cohort Study. Clin Chem. 2025 Sep 3;71(9):993-1004. doi: 10.1093/clinchem/hvaf066. PMID 40509918